CLINICAL TRIAL: NCT00316667
Title: Health2006 - an Observational Population-based Study of Cardiovascular Disease, Type 2 Diabetes, Asthma and Allergy
Brief Title: Health2006 - an Observational Study of Cardiovascular Disease, Diabetes, Asthma and Allergy
Status: Completed | Type: Observational
Sponsor: Glostrup University Hospital, Copenhagen (Other)
Collaborators: Steno Diabetes Center Copenhagen (Other)
Responsible Party: Principal Investigator, Allan Linneberg, Research Manager, Glostrup University Hospital, Copenhagen
Other Study IDs: KA20060011
Record Dates: First submitted 2006-04-19; First posted 2006-04-21 (Estimated); Last update posted 2012-10-03 (Estimated); Status verified 2012-10

CONDITIONS: Cardiovascular Disease; Type 2 Diabetes; Asthma; Hypersensitivity; Osteoporosis
Keywords: epidemiology; risk factors
MeSH Terms: conditions — Cardiovascular Diseases; Diabetes Mellitus, Type 2; Asthma; Hypersensitivity; Osteoporosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Extracted DNA, urine, serum

SUMMARY:
The aim is to assess the population prevalence of risk factors for different chronic diseases such as cardiovascular disease, type 2 diabetes, osteoporosis, asthma, and allergy. Risk factors include genetic and serologic biomarkers, questionnaire data on health and lifestyle. There are many hypotheses under study for each research field.

DETAILED DESCRIPTION:
A population-based random sample of persons living in Copenhagen is drawn from the Danish Civil Registration System and invited for a health examination including blood sample drawing, measurement of lung function, serologic and genetic biomarkers, questionnaires on lifestyle and health. The study will form the basis for research within many different areas such as cardiovascular disease, type 2 diabetes, asthma, and allergy.

ELIGIBILITY:
Inclusion Criteria:

* Persons living in 11 municipalities in Copenhagen

Exclusion Criteria:

* Pregnancy
* Non-Danish citizenship

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Random sample of citizens living in 11 municipalities in Copenhagen. Age 18-69 years.
Sampling Method: Probability Sample
Enrollment: 3471 (Actual)
Dates: Start 2006-06; Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Allan Linneberg, MD, PhD, Principal Investigator — Glostrup University Hospital, Copenhagen
Locations (1):
- Research Centre for Prevention and Health, Copenhagen, Glostrup, Denmark

REFERENCES:
- [Derived] Svendstrup M, Allin KH, Angquist L, Schnohr P, Jensen GB, Linneberg A, Thuesen B, Astrup A, Saris WHM, Vestergaard H, Sorensen TIA. Is abdominal obesity at baseline influencing weight changes in observational studies and during weight loss interventions? Am J Clin Nutr. 2018 Nov 1;108(5):913-921. doi: 10.1093/ajcn/nqy187. PMID 30475965
- [Derived] Ahluwalia TS, Troelsen JT, Balslev-Harder M, Bork-Jensen J, Thuesen BH, Cerqueira C, Linneberg A, Grarup N, Pedersen O, Hansen T, Dalgaard LT. Carriers of a VEGFA enhancer polymorphism selectively binding CHOP/DDIT3 are predisposed to increased circulating levels of thyroid-stimulating hormone. J Med Genet. 2017 Mar;54(3):166-175. doi: 10.1136/jmedgenet-2016-104084. Epub 2016 Sep 14. PMID 27627987